CLINICAL TRIAL: NCT05351671
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Dose Range Finding Study to Assess the Safety, Tolerability, PD and PK of RLS-0071 in Healthy Adult Subjects After Challenge With Inhaled Lipopolysaccharide (LPS)
Brief Title: A Clinical Study to Determine the Safety, Tolerability and Effect of RLS-0071 Doses When Given to Healthy Adults After Inhaling LPS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReAlta Life Sciences, Inc. (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLS-0071-103; 2021-006288-26 (EudraCT Number)
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — RLS-0071

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated to either of the treatment arms with RLS-0071 or the placebo arm in a 1:1:1 ratio. Subjects will be permitted to participate in only 1 arm of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the entire study, subjects, Investigators, the Sponsor, and all other persons involved in the conduct of the study will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A (Experimental): RLS-0071 lower dose group
  Interventions: Drug: RLS-0071 (10 mg/kg intravenously every 8 hours for total of 3 doses)
- Arm B (Experimental): RLS-0071 higher dose group
  Interventions: Drug: RLS-0071 (loading dose of 120 mg/kg followed by 40 mg/kg every 8 hours for 2 additional doses)
- Arm C (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo (saline dosed every 8 hours for a total of 3 doses)

INTERVENTIONS:
Drug: RLS-0071 (10 mg/kg intravenously every 8 hours for total of 3 doses) — After challenge with inhaled LPS, subjects will receive IV infusion of RLS-0071 at 10 mg/kg every 8 hours for total of 3 doses.
  Arms: Arm A
Drug: RLS-0071 (loading dose of 120 mg/kg followed by 40 mg/kg every 8 hours for 2 additional doses) — After challenge with inhaled LPS, subjects will receive IV infusion of RLS-0071 at a loading dose of 120 mg/kg followed by 40 mg/kg every 8 hours for 2 additional doses.
  Arms: Arm B
Drug: Placebo (saline dosed every 8 hours for a total of 3 doses) — After challenge with inhaled LPS, subjects will receive IV infusion of placebo (saline) dosed every 8 hours for a total of 3 doses.
  Arms: Arm C

SUMMARY:
This is a Phase 1b, randomized, double-blind, placebo-controlled, dose range finding study to assess the safety, tolerability, pharmacodynamics (PK) and pharmacokinetics (PD) of RLS-0071 in healthy adult subjects after challenge with inhaled lipopolysaccharide (LPS).

Clinical data are required to determine the potential benefit of RLS-0071, a novel drug that specifically inhibits multiple inflammatory pathways, for the treatment of severe asthma. This study has been designed to evaluate the efficacy of IV administered RLS-0071 to reduce inflammation symptoms in healthy subjects challenged with inhaled LPS, a well-known agent that produces a safe and well-controlled inflammatory response in the lung. This is a critical proof-of-concept study and dose-optimization study for future studies in severe asthma patients.

A total of 48 healthy adult subjects are planned to be enrolled in this study. Subjects will be randomly allocated to either of the treatment arms (Arm A or Arm B) with RLS-0071 or the placebo arm (Arm C) in a 1:1:1 ratio. Subjects will either receive intravenous infusion of RLS-0071 at a lower dose every 8 hours for a total of 3 doses (Arm A), RLS-0071 at a higher dose every 8 hours for a total of 3 doses (Arm B) or placebo dosed every 8 hours for a total of 3 doses (Arm C). Each subject completing the study will be evaluated for up to a total of 7 days. Subjects will be permitted to participate in only 1 arm of the study. Subjects discontinuing the study before data was collected at 6 hours post LPS challenge will be considered dropouts and will be replaced.

DETAILED DESCRIPTION:
The inclusion of a double-blind design allows a comparison between subjects receiving RLS-0071 and placebo subjects who are experiencing the same procedures and restrictions in an unbiased manner. The inclusion of a placebo control group will facilitate the distinction between efficacy signals and possible procedural/environmental events.

Eligibility criteria have been included to mitigate the risk to study subjects. Vulnerable populations such as children are excluded, as well as subjects whose medical history suggest a higher risk of experiencing adverse effects.

LPS inhalation is used in this study to be able to evaluate proof-of-concept efficacy of RLS-0071 in otherwise healthy subjects. Thus, PD assessments will be conducted to provide evidence of target engagement and guide the design of future severe asthma studies.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 to 55 years, inclusive, at the time of Screening
2. Female subjects of childbearing potential must agree to use a highly effective contraceptive method from Screening until 30 days after the last investigational medicinal product (IMP) intake and have a negative pregnancy test at Screening (blood test). The following contraceptive measures can achieve a failure rate of less than 1% per year when used consistently and correctly and are considered highly effective measures:

   1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral / intravaginal / transdermal)
   2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral / injectable / implantable)
   3. intrauterine device
   4. intrauterine hormone-releasing system
   5. bilateral tubal occlusion
   6. vasectomized partner (provided that the partner is the sole sexual partner of the woman of childbearing potential and has received medical assessment of the surgical success)
   7. sexual abstinence (only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment). Abstinence is only accepted as true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods and withdrawal] is not an acceptable method of contraception).

   Female subjects who are not of childbearing potential are exempt from contraceptive requirements. To be considered of non-childbearing potential female subjects must meet the following requirements: Must be permanently sterile (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at least 3 months before first dosing with the investigational medicinal product) or postmenopausal (defined as no menses for 12 months without an alternative medical cause).
3. A male study subject must agree to use a double barrier method (eg, condom and spermicide) during sexual contact with a pregnant woman or a woman of childbearing potential ,and agree to not donate sperm during the study and for at least 90 days after the last dose of the IMP
4. Medically healthy on the basis of medical history, physical examination, and clinical laboratory testing in the opinion of the Investigator
5. Nonsmokers and nonusers of nicotine-containing products, including vaping devices for at least 6 continuous months before the first dosing with the investigational medicinal product and for the duration of the study, to be confirmed by cotinine testing at Screening and a smoking history of < 5 pack years
6. Negative alcohol testing at Screening and Day 1
7. Negative cotinine and drug screen testing at Screening.
8. Vital signs (after semi-recumbent for at least 5 minutes) that are within the following ranges at Screening:

   1. Systolic blood pressure (BP): 90 to 140 mmHg, inclusive
   2. Diastolic BP: 50 to 90 mmHg, inclusive
   3. HR: > 45 to ≤ 100 bpm
9. Weight ≤ 100 kg and body mass index ≥ 18 and ≤ 32 kg/m2 at Screening
10. Normal renal function, defined as estimated creatinine clearance > 90 mL/min at Screening; an Investigator can determine based on clinical judgment whether a lower clearance rate can be accepted based on the muscle composition of the subject
11. Willing and able to understand the information on the nature, the scope, and the relevance of the clinical study, and to provide voluntary, written informed consent to participate in the study
12. Able to communicate well with the Investigator and/or study site personnel and to comply with the requirements of the entire study

Exclusion Criteria:

1. Use of any prescription or over-the-counter (OTC) medications, herbal products (eg, cannabidiol, St John's Wort, milk thistle), or supplements/vitamins within 14 days or 5 half-lives (whichever is longer) before first dosing with IMP and for the duration of the study, with the exception of those approved by the Investigator and Sponsor (eg, oral contraceptives, hormone replacement therapy, acetaminophen for pain relief).
2. Receipt of any investigational agent or treatment within 30 days or 5 half-lives, whichever is longer, before first dosing with IMP, or concurrent participation in another clinical study.
3. Receipt of any protein- or antibody-based therapeutic agents (eg, growth hormones or monoclonal antibodies) within 3 months before first dosing with IMP.

   Note: Influenza and COVID-19 vaccines will be allowed if all doses in the regimen have been administered more than 21 days before first dosing with IMP.
4. History of any major surgery within 6 months before first dosing with IMP.
5. Prior diagnosis of COVID 19 within 90 days before first dosing with IMP.
6. History of hepatic disease, or current clinically significant liver function test results, defined as ALT, AST, total bilirubin and fractionated bilirubin, or alkaline phosphatase > 1.5 × upper limit of normal (ULN) at Screening.

   Note: Isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated, and direct bilirubin is < 35%.
7. History of any clinically relevant or chronic psychiatric, renal, hepatic, pancreatic, cardiovascular, neurological, hematological, or gastrointestinal abnormality (eg, inflammatory bowel disease)
8. History of severe allergic/anaphylactic reaction
9. History of autoimmune disease including glomerulonephritis
10. Known hypersensitivity to the active substance or to any of the excipients of each IMP including lipopolysaccharide (LPS) and polyethylene glycol (PEG)
11. History of any active infection within 14 days before dosing with IMP, if deemed clinically significant by the Investigator and Sponsor
12. Any acute illness within 30 days before dosing with IMP
13. Lower respiratory tract infection within 3 months before first dosing with IMP
14. History of warfarin use or International Normalized Ratio ≥ 1.5
15. History (within 2 years before the first dosing with IMP) of moderate or severe use disorder for any substance other than caffeine (based on the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition criteria)
16. Known diagnosis or active infection with Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV)-1 or HIV-2
17. Existence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the absorption, distribution, metabolism, or excretion of RLS-0071
18. Presence of clinically significant ECG finding (confirmed upon repeat testing) that, in the opinion of the Investigator and/or Sponsor, may interfere with any aspect of study conduct or interpretation of results
19. Concurrent conditions that could interfere with safety and/or tolerability measurements, as determined by the Investigator
20. Pregnant and/or lactating
21. Inability to produce sufficient amounts of induced sputum at baseline visit
22. Inability to tolerate IV administration
23. Poor venous access, as determined by the Investigator
24. Unable or unwilling to cooperate with the study site staff for any reason
25. Employees of the Sponsor or subjects who are employees or relatives of the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in absolute neutrophil count in induced sputum | At 6 and 24 hours after inhaled lipopolysaccharide (LPS).
  Primary PD

SECONDARY OUTCOMES:
Change from Baseline in cytokines (Th1 and Th17) in induced sputum | At 6 and 24 hours after inhaled LPS.
  Secondary PD

OTHER OUTCOMES:
Change from Baseline in MPO level in sputum | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
Change from Baseline in concentration of myeloperoxidase (MPO) binding in blood | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
Change from Baseline in amount of cell-free DNA in blood. | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
Change from Baseline in C-reactive protein in blood | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
Change from Baseline in interleukin (IL)-6 in exhaled breath particles. | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
Change from Baseline in peripheral absolute neutrophil count in blood | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
Change from Baseline in neutrophil percentage in sputum | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
RLS-0071 concentration in induced sputum | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
Change from Baseline in complement activity assay immune-complex membrane attack complex [IC-MAC] in blood. | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
Change from Baseline in complement activity assay immune-complex membrane attack complex [IC-MAC] in sputum. | At 6 and 24 hours after inhaled LPS.
  Exploratory PD
Cmax of RLS-0071 | Days 1 and 2, 5 minutes after completing each infusion of study treatment
  Exploratory PK
Frequency and severity of treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs) and deaths | Day 1 - start of treatment, Day 2 - end of treatment, and through Day 7 - end of study visit
  Safety endpoint
Frequency of premature discontinuation of the investigational medicinal product (IMP) due to TEAEs | Day 1 - start of treatment, Day 2 - end of treatment, and through Day 7 - end of study visit
  Safety endpoint
Change from Baseline in Complete Blood Count (CBC) | Day minus 6 through Day 7 at end of study
  Safety endpoint
Vitals sign - blood pressure | Day minus 29 through Day 7 at end of study
  Safety endpoint
Vitals sign - weight | Day minus 29 through Day 7 at end of study
  Safety endpoint
Vitals sign - renal function (estimated creatinine clearance) | Day minus 29 through Day 7 at end of study
  Safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Cunnion, MD, MPH, Study Chair — ReAlta Life Sciences, Inc.; Linda Dell, Study Director — ReAlta Life Sciences, Inc.
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine (ITEM), Hanover, Germany